CLINICAL TRIAL: NCT05525949
Title: Treatment of Homonymous Visual Loss With Digital Therapeutics, VIVID Brain, Visual Perceptual Learning Device (HOGWAND Trial) : Multi Center, Randomized, Single-blind (Evaluator), Superiority Prove, Prospective Confirmatory Trial
Brief Title: Visual Perceptual Learning Based Digital Therapeutics for Visual Field Defect After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nunaps Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NNS-VB-02
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-12

CONDITIONS: Visual Fields Hemianopsia; Hemianopsia, Homonymous
Keywords: Visual field defect; Visual perceptual learning; Humphrey visual field
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIVID Brain (Experimental): VIVID Brain, 5 times a week for 12 weeks
  Interventions: Device: VIVID Brain
- No-treatment Control (Other): No-treatment is administered during control period.
  Interventions: Other: No-treatment Control

INTERVENTIONS:
Device: VIVID Brain — Participants receive visual perceptual training using the VIVID Brain software.
  Arms: VIVID Brain
Other: No-treatment Control — No-treatment is administered during control period.
  Arms: No-treatment Control

SUMMARY:
This study evaluates the efficacy of visual perceptual learning for the treatment of visual field defect caused by brain disease. Half of participants will receive visual perceptual training using the VIVID Brain. The other half will not receive any training because there is no standard treatment for visual field defect caused by brain disease.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older
* At least 3 months after brain disease related to visual field defect
* Verified brain disease in visual pathway related to occipital lobe, parietal lobe, temporal lobe or etc. using CT or MRI
* Brain disease induced visual field defect
* Able to use the VR(Virtual Reality) device
* Able to use the app with a smart phone
* Patient/legally authorized representative has signed the informed consent form

Exclusion Criteria:

* Complete hemianopsia
* Epilepsy, photosensitivity, Parkinson's disease
* Bilateral visual field defect
* Hemispatial neglect
* Ophthalmologic disorder that may interfere the trial. (Ptosis of Eyelid, Corneal Opacity, Diabetic Retinopathy, Glaucoma, Macular Degeneration etc.)
* Inability to discontinue psychostimulants such as methylphenidate, modafinil, and amphetamine.
* Candidate for carotid endarterectomy or stenting
* Received ophthalmologic surgery or laser surgery within 3 months, except for the cataract surgery
* Pregnant or breast feeding
* Participating in other clinical trial
* Any other condition that, in the opinion of the investigator, precludes participation in the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
The sum of improved areas compared to baseline in the whole field | 12 weeks
  The sum of areas where sensitivity increased by more than 6 dB compared to baseline in the whole field measured by Humphrey visual field test.
  The improved area ranges between 0 and 2,736 degree^2, of which larger area indicates better outcome.

SECONDARY OUTCOMES:
The sum of improved areas compared to baseline in the affected hemi-field | 12 weeks
  The sum of areas where sensitivity increased by more than 6 dB compared to baseline in the affected hemi-field measured by Humphrey visual field test.
Changes in perimetric mean deviation relative to baseline in the whole field | 12 weeks
  Changes in perimetric mean deviation relative to baseline in the whole field measured by Humphrey visual field test.
Changes in mean total deviation relative to baseline in the affected hemi-field | 12 weeks
  Changes in mean total deviation relative to baseline in the affected hemi-field measured by Humphrey visual field test.

CONTACTS AND LOCATIONS:
Overall Officials: Gyeong-Moon Kim, MD, PhD, Study Chair — Samsung Medical Center
Locations (12):
- South Korea (12):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Daejeon Eulji University Medical Center, Daejeon
  - Inje University Ilsan Paik Hospital, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Namgung E, Kim BJ, Kwon JH, Han MK, Kim HY, Jung JM, Kim JG, Park KY, Koo J, Hong KS, Yu KH, Cho AH, Chang JY, Kwon SU, Lee BJ, Choi HG, Cho M, Kim GM, Kang DW. Personalized Visual Perceptual Learning Digital Therapy for Visual Field Defects Following Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2511068. doi: 10.1001/jamanetworkopen.2025.11068. PMID 40388168